CLINICAL TRIAL: NCT05452642
Title: Supporting Understanding of PCOS Education and Research. Official Title: Glycemic Reduction Approaches in Polycystic Ovary Syndrome: a Comparative Effectiveness Study
Brief Title: The Supporting Understanding of PCOS Education and Research (SUPER) Study
Acronym: SUPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00210749; 1R01DK128205-01A1 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary
Keywords: Very low carbohydrate diet; Dietary approaches to stop hypertension (DASH) diet; Nutrition therapy
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment and data analysis will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH diet (Active Comparator): 12-month DASH diet intervention with psychological support
  Interventions: Behavioral: DASH diet
- Very low-carbohydrate diet (Experimental): 12-month very low-carbohydrate diet intervention with psychological support
  Interventions: Behavioral: Very low-carbohydrate diet

INTERVENTIONS:
Behavioral: DASH diet — Participants in this arm will be taught a DASH diet plus psychological skills to support dietary adherence.
  Arms: DASH diet
Behavioral: Very low-carbohydrate diet — Participants in this arm will be taught a very low-carbohydrate diet plus psychological skills to support dietary adherence.
  Arms: Very low-carbohydrate diet

SUMMARY:
This research will test whether a Dietary Approaches to Stop Hypertension (DASH) or a very low-carbohydrate diet better improves outcomes like blood glucose control and body weight for adults with polycystic ovary syndrome.

Participants will have screening (includes blood draw) and baseline testing with a continuous glucose monitor and a body composition scan (called a dual-energy x-ray absorptiometry or DEXA). Once these enrollment steps are completed and the participants will be randomized to one of two 12-month programs.

ELIGIBILITY:
Inclusion criteria:

* Participants must have the following criteria:

  * oligomenorrhea-anovulation

    * spontaneous intermenstrual periods (if not on hormonal birth control or birth control that alters menstrual cycle timing) of < 21 days or > 35 days or a total of 8 or fewer menses per year
    * if on hormonal birth control or birth control that alters menstrual cycle timing, a history of irregular periods
  * and hyperandrogenism

    * If not on hormonal birth control or birth control that alters menstrual cycle timing: Total testosterone ≥ 35 ng/dL OR free testosterone > 4.0 pg/ml OR free androgen index > 1.5 OR in-person scoring for hirsutism, based on the modified Ferriman-Gallwey score, if attending an in-person assessment or based on the self-assessment (if not attending an in-person assessment) with a score of ≥ 4 considered hirsutism;
    * If on hormonal birth control or birth control that alters menstrual cycle timing: Tests within the past 10 years showing the above or study team's in-person assessment of hirsutism as above.
* If no medical records to confirm (most recent test from within the last 10 years in range), tests for diagnosis will be ordered:

  * total testosterone < 100 ng/dL,
  * dehydroepiandrosterone sulfate (DHEAS) < 600 μg/dL,
  * fasting 17-hydroxyprogesterone (17-OHP) level < 2.0 ng/mL,
  * prolactin < 25 ng/ml),
  * follicle-stimulating hormone (FSH) levels < 20 mIU/mL
* BMI 25-50 kg/m2 or 23-50 kg/m2 for Asians
* Access to internet
* Ability to engage in light physical activity
* Willingness to be randomized to either dietary approach
* Measured HbA1c at baseline of 5.3%-9.0%

Exclusion criteria:

* Primary

  * Patients with non-PCOS etiologies of anovulation and hyperandrogenism (Cushing's disease, thyroid dysfunction, elevated prolactin levels, signs of a congenital adrenal hyperplasia organic intracranial lesion like a pituitary tumor, or suspected adrenal or ovarian tumor secreting androgens)
  * Menopause or removal of the ovaries
  * history of type 1 diabetes
  * use of medications prescribed for weight loss or psychostimulants known to affect weight
  * participation in another weight loss program or intervention
  * use of glucose lowering medications other than metformin or medications known to affect metabolism, such as chronic oral corticosteroids
  * pregnant or planning to become pregnant during the intervention period
  * Breastfeeding or less than 6 months postpartum
  * previous bariatric surgery or planning to have bariatric surgery during the study period
  * Self-reported blood disorders that influence HbA1c, including frequent blood transfusions, phlebotomy, anemia, hemoglobinopathy, and polycythemia
* Ability

  * inability to read, write, or speak English
  * inability to provide informed consent
  * adherence to a vegan or vegetarian diet
  * difficulty chewing or swallowing
  * no influence over what foods are purchased, prepared, and/or served or inability to follow dietary advice due to lack of money or other resources
  * above weight limit (500 lbs) for DEXA
  * self-report of alcohol or substance use disorder within the past 5 years, including current at-risk drinking based on an AUDIT score of 15 or higher (but those who score a 15 or higher and have this criterion as their only reason for ineligibility may be assessed by a clinical psychologist for alcohol use disorder and if deemed to not have such a disorder would be eligible for the trial)
* Safety

  * Renal disease: BUN > 30 mg/dL or serum creatinine > 1.4 mg/dL in our screening blood tests or history of kidney stones
  * untreated eating disorder or unstable serious mental illness (such as depression (score of 20 or greater on the PHQ8), bipolar or schizophrenia with psychosis)
  * use of warfarin
  * chronic kidney disease, stage 4 or higher
  * Any other concerning values in baseline labs (we will plan to send the participant to their PCP and allow the participant to return for later enrollment if labs are no longer concerning) Examples:

    * triglycerides of 600 mg/dL or higher
    * baseline uncorrected thyroid disease: TSH < .45 mIU/ML or > 4.5 mIU/ML
    * potassium: any abnormal value
    * baseline aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times normal
  * any condition for which the study team deems participation to be unsafe or inappropriate

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 223 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 0 to 12 months
  percentage of glycosylated hemoglobin

SECONDARY OUTCOMES:
Change in percent body weight loss | 0-12 months
  percent change
Change in glycemic variability | 0 to 12 months
  This will be measured with an Abbott Libre Pro continuous glucose monitoring device on participants' upper arm and the information on the sensor is blinded to participants.
  The monitoring device will record participants' glucose levels in the interstitial fluid by a glucose oxidase method every 15 minutes, continuously for 14 days at each time point.
  The glucose variability and the proportion of time spent in the euglycemic (3-7.8 millimoles per litre (mmol/l)) and hyperglycemic (≥ 11.1 mmol/l for at least 15 minutes) states, following previous standards for interstitial glucose concentrations.
Change in percent body fat on DEXA | 0 to 12 months
  This will be measured by dual-energy X-ray absorptiometry scan
Change in HbA1c | 0 to 4 months
  percentage of glycosylated hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Laura Saslow, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Greenwell S, Jones A, Smith YR, Marriott D, Aikens JE, Padmanabhan V, Saslow LR. Protocol for a randomized comparative effectiveness trial comparing a very low-carbohydrate diet to DASH diet for polycystic ovary syndrome: the SUPER (Supporting Understanding of PCOS Education and Research) trial. Trials. 2024 Nov 9;25(1):750. doi: 10.1186/s13063-024-08583-y. PMID 39516828

DOCUMENTS (1):
  • Informed Consent Form (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT05452642/ICF_000.pdf